CLINICAL TRIAL: NCT02486692
Title: Pilot Evaluation of AboutFace: A Novel Peer Education Resource for Veterans
Brief Title: Pilot Evaluation of AboutFace: Novel Peer Education Resource for Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PPO 14-360
Record Dates: First submitted 2015-06-16; First posted 2015-07-01 (Estimated); Results first posted 2019-05-06 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-05

CONDITIONS: PTSD
Keywords: Mental Health; PTSD; Stigma; Peer Education; Web Education; Self Help
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Psychological Well-Being; Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase II- Experimental Group (Experimental): Participants were provided with instructions and a web link for accessing the AboutFace website after the baseline assessment.
  Interventions: Other: AboutFace Website
- Phase II- Usual Care Group (No Intervention): Participants were provided with instructions and a web link for accessing some online PTSD education materials after the baseline assessment.

INTERVENTIONS:
Other: AboutFace Website — AboutFace is an informational website that utilizes digital storytelling to describe PTSD symptoms and different treatments for PTSD.
  Arms: Phase II- Experimental Group

SUMMARY:
The purpose of this study is to evaluate the AboutFace peer education website for the purpose of reducing stigma and improving attitudes toward seeking mental health services among Veterans.

DETAILED DESCRIPTION:
Research suggests that at least 1 in 10 Veterans will meet criteria for posttraumatic stress disorder (PTSD) related to their military experience. Treatment is widely available to Veterans with PTSD, and national dissemination initiatives have increased Veterans' access to best practice interventions. However, treatment seeking remains strikingly low among Veterans with PTSD. In fact, most Veterans with PTSD do not seek mental health services due to perceived stigma and other associated barriers. The National Center for PTSD recently developed and launched AboutFace, a peer education resource for Veterans. The investigators of this study believe that AboutFace has tremendous potential to reduce stigma and improve attitudes toward seeking mental health services among Veterans. However, it has not yet been evaluated. Investigators have partnered with the National Center for PTSD to launch this mixed methods pilot evaluation of AboutFace. There will be two phases to this study. During Phase I- Usability, 20 Veterans will be recruited to participate in individual interviews during which they will be asked to describe the ease of use of the AboutFace website for the researchers. During Phase II- Feasibility, 60 Veterans will be randomized to one of two conditions- About Face or Usual Care. All participants will complete several brief assessments measuring PTSD symptoms and attitudes toward seeking mental health services. Participants will then be randomized to either receive a link to the About Face website or to receive a link to a general online brochure about PTSD. After two weeks, participants will complete the assessment measures once again to determine any changes in attitudes toward seeking mental health services and potential changes in PTSD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age
* Recommended for PTSD treatment following evaluation
* Internet access
* English Speaking

Exclusion Criteria:

* Minors under the age of 18
* Non-Veterans
* Negative for PTSD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-04; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J Ruggiero, PhD MA BA, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kreuze E, Jenkins C, Gregoski M, York J, Mueller M, Lamis DA, Ruggiero KJ. Technology-enhanced suicide prevention interventions: A systematic review. J Telemed Telecare. 2017 Jul;23(6):605-617. doi: 10.1177/1357633X16657928. Epub 2016 Jul 3. PMID 27377792
- [Derived] Hamblen JL, Grubaugh AL, Davidson TM, Borkman AL, Bunnell BE, Ruggiero KJ. An Online Peer Educational Campaign to Reduce Stigma and Improve Help Seeking in Veterans with Posttraumatic Stress Disorder. Telemed J E Health. 2019 Jan;25(1):41-47. doi: 10.1089/tmj.2017.0305. Epub 2018 May 10. PMID 29746232
- [Derived] Bunnell BE, Davidson TM, Hamblen JL, Cook DL, Grubaugh AL, Lozano BE, Tuerk PW, Ruggiero KJ. Protocol for the evaluation of a digital storytelling approach to address stigma and improve readiness to seek services among veterans. Pilot Feasibility Stud. 2017 Feb 17;3:7. doi: 10.1186/s40814-017-0121-3. eCollection 2017. PMID 28239485

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase II-Experimental: Participants using AboutFace
  AboutFace Website: AboutFace is an informational website that utilizes digital storytelling to describe PTSD symptoms and treatment for PTSD.
- Phase II- Usual Care Condition: Education and Print materials only
Period: Overall Study
Arm/Group | Phase II-Experimental | Phase II- Usual Care Condition
Started | 30 | 30
Completed | 26 | 23
Not Completed | 4 | 7
Not completed — did not login for randomization | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase II-Experimental | Phase II- Usual Care Condition | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 27 | 55
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Full Range); unit: years] | 42.27 [18 to 80] | 42.13 [18 to 69] | 42.20 [18 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 19 | 24 | 43
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Endorsed and Anticipated Stigma Inventory (EASI)
Description: THE EASI assesses for perceptions of treatment effectiveness, stigma, and external barriers to treatment seeking. Answers are ranked from 1 to 5 with 1 being "Strongly Disagree" and 5 being "Strongly Agree" and higher scores are indicative of greater stigma. Total scores can range from 40 to 190.
  Phase I participants did not participate in Phase II (the clinical trial portion of the study) and were not assessed using this measure.
Time Frame: pre-treatment (baseline) & post-treatment (two-week) assessment
Population: Total N=60; Only 49 randomized (26 in EXP arm and 23 in Usual Care arm) because 11 participants did not access website portal to obtain their randomization assignment. The EASI was also missing for 1 participant at post.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase II-Experimental | Phase II- Usual Care Condition
Number analyzed (Participants) | 26 | 22
units on a scale
  pre-treatment (baseline) mean | 57.9 (27.2) | 62.3 (31.4)
  post-treatment (2-week) mean | 57.5 (33.1) | 54.1 (30.7)

2. Primary Outcome: PTSD Checklist (PCL-V)
Description: The PCL-V is a 20-item self-report measure that assesses PTSD severity. Individual item responses can range from 0-4 with 0 being "Not At All" and 4 being "Extremely" and total scores can range from 0 to 80. Higher numbers on the PCL-V are indicative of greater PTSD severity.
  Phase I participants did not participate in Phase II (the clinical trial portion of the study) and were not assessed using this measure.
Time Frame: pre-treatment (baseline) & post-treatment (2-week) assessment
Population: Total N=60; Only 49 randomized (26 in EXP arm and 23 in Usual Care arm) because 11 participants did not access the website portal to obtain their randomization assignment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase II-Experimental | Phase II- Usual Care Condition
Number analyzed (Participants) | 26 | 23
units on a scale
  pre-treatment (baseline) mean (sd) | 51.1 (10.6) | 52.1 (11.4)
  post-treatment (2-week) mean (sd) | 49.4 (9.7) | 49.5 (12.5)

3. Primary Outcome: PTSD Treatment Initiators
Description: percentage/rate of PTSD treatment initiation at post assessment (2-weeks) Phase I participants did not participate in Phase II (the clinical trial portion of the study) and were not assessed using this measure.
Time Frame: two weeks post assessment
Population: Total N=60; Only 49 randomized (26 in EXP arm and 23 in Usual Care arm) because 11 participants did not access the website portal to obtain their randomization assignment. Data was also missing for 1 participant at post.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II-Experimental | Phase II- Usual Care Condition
Number analyzed (Participants) | 26 | 22
Participants | 20 | 15

ADVERSE EVENTS:
Time Frame: Up to two weeks for Phase II participants (baseline to 2 weeks post assessment).
Description: No adverse events were reported in Phase I. Participation involved a single visit.
Groups:
- Phase II- Experimental: Participants using AboutFace
  AboutFace Website: AboutFace is an informational website that utilizes digital storytelling to describe PTSD symptoms and treatment for PTSD.
Arm/Group | Phase II- Experimental | Phase II- Usual Care Condition
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No